CLINICAL TRIAL: NCT07236255
Title: The Effect of Education Provided Using Video and Podcast Applications Developed With the Health Action Process Approach Model on Breastfeeding Self-Efficacy and Breastfeeding Success in Primiparous Mothers: A Mixed Study
Brief Title: The Effect of Model-based Education on Breastfeeding Self-efficacy and Success
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Yalcin (Other)
Responsible Party: Sponsor-Investigator, Esra Yalcin, Lecturer, Bozok University
Organization: Bozok University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBF-EY-2323
Record Dates: First submitted 2025-11-16; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Primiparous Pregnant Women in the Third Trimester
Keywords: breastfeeding self-efficacy; podcast; breastfeeding success; video; primiparous pregnant women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): To administer the pre-test, pregnant women will complete the Introductory Information Form, the Breastfeeding Attitudes Assessment Scale, and the Breastfeeding Self-Efficacy Scale-Short Form. After completing the questionnaires, they will receive breastfeeding education and a video and podcast created by the researcher based on the Health Action Process Approach Model. Pregnant women will be contacted on the day of delivery and asked to re-watch the video and listen to the podcast. One month postpartum, pregnant women will complete the Breastfeeding Attitudes Assessment Scale, the Breastfeeding Self-Efficacy Scale-Short Form, the LATCH Breastfeeding Diagnosis and Assessment Scale, and the Breastfeeding Follow-up Form I. A post-test will be administered at six months, and they will complete the Breastfeeding Attitudes Assessment Scale, the Breastfeeding Self-Efficacy Scale-Short Form, the LATCH Breastfeeding Diagnosis and Assessment Scale, and the Breastfeeding Follow-up Form II.
  Interventions: Behavioral: Breastfeeding Education
- control group (No Intervention): To administer the pretest, pregnant women will complete the Introductory Information Form, the Breastfeeding Attitudes Assessment Scale, and the Breastfeeding Self-Efficacy Scale-Short Form. After completing the questionnaires, they will be provided with a Breastfeeding Brochure from the Turkish Ministry of Health. One month after birth, pregnant women will complete the Breastfeeding Attitudes Assessment Scale, the Breastfeeding Self-Efficacy Scale-Short Form, the LATCH Breastfeeding Diagnosis and Assessment Scale, and the Breastfeeding Follow-up Form I. A posttest will be administered at six months, and pregnant women will complete the Breastfeeding Attitudes Assessment Scale, the Breastfeeding Self-Efficacy Scale-Short Form, the LATCH Breastfeeding Diagnosis and Assessment Scale, and the Breastfeeding Follow-up Form II.

INTERVENTIONS:
Behavioral: Breastfeeding Education — Before the intervention, interviews will be conducted with pregnant women based on the Health Action Process Approach Model to identify any deficiencies related to breastfeeding. As a result, videos and podcasts based on the model will be produced. The intervention group will receive breastfeeding education, distribute these videos and podcasts, and be asked to watch them. Pregnant women will be contacted after birth to provide reminders. The control group will not receive any interventions and will only receive the breastfeeding guidelines from the Turkish Ministry of Health.
  Arms: experimental group

SUMMARY:
This study was designed as a randomised, pretest-posttest study, assessing breastfeeding self-efficacy and breastfeeding in first-time mothers following a separate video and podcast training session using the Health Action Process Approach Model. The study will be conducted with primiparous pregnant women in their third trimester, with no restrictions on breastfeeding. In the first phase of the study, a semi-trained interview format based on the SESY Model will be administered to 15 pregnant women at a fertility school to address nutritional deficiencies. Deficiencies in the pregnant women will be identified. To address these deficiencies, the researcher will develop a breastfeeding education book based on the SESY Model, produce a video, and produce the same content as a podcast. Both groups will complete the Introductory Information Form, the Breastfeeding Attitudes Assessment Scale, and the Breastfeeding Self-Efficacy Scale-Short Form. After completing their surveys, the control groups, which are pregnant women, will only receive the Breastfeeding Brochure from the Ministry of Health of the Republic of Turkey. Pregnant women in the intervention groups receive breastfeeding education throughout the cycle, in addition to videos and podcasts. Pregnant women will be asked to watch the videos and listen to the podcast until they give birth. Pregnant women will be contacted on the day of their birth to ask if there are any websites they would like to learn more about and to re-watch the video and listen to the podcast. Pregnant women will be contacted for an evaluation one month after birth to complete the Breastfeeding Attitudes Assessment Scale, Breastfeeding Self-Efficacy Scale-Short Form, LATCH Breastfeeding Diagnostic and Assessment Scale, and Breastfeeding Follow-Up Form I. To emphasize the importance of breastfeeding in the first six months and ensure continuity of breastfeeding, pregnant women will be contacted again at six months to complete a post-test and the Breastfeeding Attitudes Assessment Scale, Breastfeeding Self-Efficacy Scale-Short Form, LATCH Breastfeeding Diagnostic and Assessment Scale, and Breastfeeding Follow-Up Form II.

DETAILED DESCRIPTION:
This study was designed as a phenomenological, randomized, pretest-posttest study to measure breastfeeding self-efficacy and breastfeeding success in first-time mothers following education delivered using a separate video and podcast application using the Health Action Process Approach Model. The study will be conducted in a maternity school and a breastfeeding room at a hospital in Türkiye. The research population will consist of all pregnant women who pay their dues to the hospital's maternity clinic. The sample will consist of primiparous pregnant women who refuse to participate, have no communication problems in Turkish, have at least a primary school education, are in a healthy pregnancy, are scheduled for vaginal or cesarean delivery, are in their third trimester, and have no breastfeeding restrictions. In the first phase of the study, a semi-trained interview format based on the SESY Model will be administered to 15 pregnant women at the reproductive school to address their breastfeeding needs. During the session, any distractions (clocks, pictures, charts, etc.) in the room will be removed. To prevent interruptions during the interview, a warning message will be sent to the door, and the pregnant woman will be asked to silence her phone. Care will be taken to maintain a conversational tone, allowing the pregnant woman to express herself freely. Information about the interview duration will be provided at the pregnant woman's request. The interview will last approximately 15-20 minutes. The interview will examine pregnant women's knowledge of breastfeeding, their attitudes toward breastfeeding, their expectations, potential problems, breastfeeding concerns, and their focus on these issues. Deficiencies in the pregnant women will be identified. Content analysis and descriptive analysis will be used to identify breastfeeding-related solutions and identify the appropriate training locations. Due to these deficiencies, the researcher will prepare a breastfeeding education booklet based on the SESY model, produce a video, and the same content will be produced as a podcast. Experts will be consulted on the content before and after the video and podcast are produced. The appropriate order of the opinions will be determined by the video and podcast, while the control group will only use the Breastfeeding Brochure from the Ministry of Health of the Republic of Turkey. To record the test, pregnant women in both the intervention and control groups will be contacted and invited to the hospital conference room. Both groups will complete the Introductory Information Form, the Breastfeeding Attitudes Assessment Scale, and the Breastfeeding Self-Efficacy Scale-Short Form. After completing the questionnaires, pregnant women in the control groups will only receive the Breastfeeding Brochure from the Ministry of Health of the Republic of Turkey. Pregnant women in the intervention group will receive breastfeeding education at the school, along with videos and podcasts. Pregnant women will be asked to watch the video and listen to the podcast until delivery. On the day of delivery, pregnant women will be contacted to ask if there are any sites where they would like to receive information and will be asked to rewatch the video and listen to the podcast. Pregnant women will be contacted for an evaluation at the first month postpartum and will complete the Breastfeeding Attitudes Assessment Scale, the Breastfeeding Self-Efficacy Scale-Short Form, the LATCH Breastfeeding Diagnostic and Assessment Scale, and the Breastfeeding Follow-up Form I. In order to ensure the importance of breast milk and the continuity of breastfeeding in the first 6 months, pregnant women will be contacted again in the 6th month to complete the post-test and Breastfeeding Attitude Measurement Assessment, Breastfeeding Self-Efficacy Scale-Short Form, LATCH Breastfeeding Diagnosis and Assessment Scale and Breastfeeding Follow-up Form II.

ELIGIBILITY:
Inclusion Criteria:

* Those who have no communication problems in Turkish
* Have at least a primary school degree
* Have a healthy pregnancy
* Are planning a vaginal or cesarean delivery
* Are in their third trimester
* Have no breastfeeding restrictions
* Are primiparous

Exclusion Criteria:

* Pregnant women who: • Are foreign nationals

  * Refuse to participate in the study
  * Have a high-risk pregnancy
  * Have vision or hearing problems
  * Have a low-birth-weight baby
  * Have a premature birth
  * Have multiple births
  * Have babies incubated after birth
  * Have a chronic disease will not be included in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Primiparous pregnant women in their third trimester
Enrollment: 100 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Attitude Assessment Scale (BATAS) | Pre-test: before the intervention, post-test after the intervention at 1 month postpartum and 6 months postpartum
  The Breastfeeding Attitude Assessment Scale was developed by Arslan in 1997. The scale aims to measure breastfeeding attitudes in mothers who have given birth. The 46-item scale is a 5-point Likert-type scale. It includes 22 positive and 24 negative breastfeeding attitude items. Positive items are scored as "Strongly Agree" (4), "Agree" (3), "Undecided" (2), "Slightly Agree" (1), and "Strongly Disagree" (0), while negative items are scored as "Strongly Agree" (0), "Agree" (1), "Undecided" (2), "Slightly Agree" (3), and "Strongly Disagree" (4). The highest possible score is 184. A high score indicates that mothers have positive attitudes toward breastfeeding. In validity and reliability studies conducted on the scale, Cronbach's alpha was calculated as 0.63.
Breastfeeding Self-Efficacy Scale-Short Form | Pre-test: before the intervention, post-test after the intervention at 1 month postpartum and 6 months postpartum
  The Breastfeeding Self-Efficacy Scale (BSS) was developed by Dennis in 1999 to assess mothers' breastfeeding self-efficacy levels. The first form consisted of 33 items. In 2003, Dennis removed some items to create a new 14-item "Breastfeeding Self-Efficacy Scale Short Form." It consists of a 5-point Likert-type scale. The lowest possible score is 14, while the highest is 70. Scoring is as follows: "Not at all sure (1)," "Not very sure (2)," "Sometimes sure (3)," "I'm sure (4)," and "Always sure (5)." Higher scores indicate higher breastfeeding self-efficacy. The Turkish validity and reliability of the short form of the scale was conducted by Aluş-Tokat and Okumuş in 2009. The Cronbach's alpha value for the Turkish version of the Antenatal Breastfeeding Self-Efficacy Scale was found to be 0.87. The Cronbach's alpha value for the Turkish version of the Postpartum Breastfeeding Self-Efficacy Scale was found to be 0.86.

OTHER OUTCOMES:
LATCH Breastfeeding Diagnostic and Assessment Scale | after intervention: 1st and 6th months postpartum
  The LATCH breastfeeding diagnosis and assessment scale is a diagnostic method used to assess breastfeeding success, first developed in 1986 using a scoring method similar to the APGAR scoring system. This measurement tool was developed to objectively diagnose breastfeeding, identify breastfeeding problems, establish a common language among healthcare professionals, and be used in research. It consists of five assessment criteria: L (latch on the breast), A (audible swallowing), T (type of nipple), C (comfort breast/nipple), and H (hold/help). Each item is scored between 0 and 2. The maximum total score is 10, with a higher score indicating higher breastfeeding success. A Turkish reliability study of the instrument was conducted by Yenal and Okumuş. The Cronbach's alpha value for the original version of the scale was 0.93, while it was found to be 0.95 in the Turkish adaptation study.
SESY-Based Breastfeeding Tracking Form I (Month 1) | after intervention: 1st and 6th months postpartum
  Breastfeeding Follow-up Form I, prepared by the researcher in line with the literature (Yılmaz, 2014; Avcı, 2024; Arslan, 2020; Köprülü, 2024), was created to evaluate breastfeeding success and monitor the babies' breastfeeding status by contacting individuals in the intervention and control groups at the first month. The form, consisting of 27 questions, assessed the mother's continued breastfeeding status.
SESY-Based Breastfeeding Tracking Form II (6th Month) | after intervention: 1st and 6th months postpartum
  The Breastfeeding Follow-up Form II, prepared by the researcher in line with the literature (Yılmaz, 2014; Avcı, 2024; Arslan, 2020; Köprülü, 2024), was created to monitor breastfeeding continuity by contacting individuals in the intervention and control groups at six months. The 28-question form inquired about the mother's breastfeeding continuity, the initiation of complementary feeding, support systems, and starting work.

IPD SHARING:
Plan to Share IPD: No
To protect participant confidentiality and because data is collected only for this study, individual participant data will not be collected.